CLINICAL TRIAL: NCT01854463
Title: The Effect of Vitamin D Supplementation on the Glycemic Control and Non-alcoholic Fatty Liver Disease in Type 2 Diabetes
Brief Title: The Effect of Vitamin D Supplementation in Type 2 Diabetes
Acronym: VD2000
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Collaborators: Korean Diabetes Association (Other)
Responsible Party: Principal Investigator, OHKHYUN RYU, Assistant Professor, Chuncheon Sacred Heart Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSHH2011-64; KDA2010 (Other Grant/Funding Number: Korean Diabetes Association year 2010 grant)
Record Dates: First submitted 2013-04-19; First posted 2013-05-15 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2013-05

CONDITIONS: DIABETES MELLITUS
Keywords: DIABETES MELLITUS; VITAMIN D; ARTERIAL STIFFNESS; FATTY LIVER; BONE TURNOVER
MeSH Terms: conditions — Diabetes Mellitus; Fatty Liver | interventions — Cholecalciferol; Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D3 (Experimental): 25-hydroxy vitamin d 2000 IU and elemeental calcium 200mg daily for 24 weeks
  Interventions: Drug: Vitamin D3
- placebo (Placebo Comparator): administered elemental calcium 200mg daily for 24 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Vitamin D3 — 2000IU per day
  Other Names: dicamax d
  Arms: Vitamin D3
Drug: placebo — elemental calcium 200mg per day per 24 weeks
  Other Names: calcium
  Arms: placebo

SUMMARY:
In many observational studies, vitamin D deficiency is related to glucose intolerance and diabetes. But there little randomized, controlled interventional studies that evaluate the effect of vitamin D in type 2 diabetes.

Investigators investigate the effect of high dose (2000IU) 25-hydroxy vitamin D on type 2 diabetes in glycemic controls, non-alcholic fatty liver disease, and arterial stiffness, and bone turnover markers.

DETAILED DESCRIPTION:
After informed consent, investigators randomized 180 type 2 diabetes into interventiona group (25-hydroxy vitamin d 2000 IU+ elemental calcium 200mg per day) or placebo group (elemental calcium 200mg per day). The participants should control diabetes by oral medications or lifestyle intervention at the intervention period. Investigators exclude the participants who took vitamin D or calcium or anti-osteoporotic drugs. Investigators also exclude renal insufficiency (Cr>1.5 in men or Cr>1.4 in women) or heavy alcoholics.

Investigators followed the participants for 24 weeks. After randomization, investigators checked HbA1c,glucose, calcium, 25-hydroxyvitamin d, AST, ALT,Creatinine, Parathyroid hormone, bone-specific alkaline phosphatase, serum CTX, brachial-ankle pulse wave velocity, central blood pressure, and aortic augmentation index, and precontrast liver computed tomography. Also investigators checked body weight, height, and peripheral blood pressure.

At 12 weeks, investigators checked HbA1c, 25-hydroxy vitamin D, AST, ALT, calcium, and creatinine.

At the end of the study(at 24 weeks), investigators checked HbA1c, glucose, AST, ALT, Creatinine, calcium, bone-specific alkaline phosphatase, serum CTX, brachial-ankle pulse wave velocity, central blood pressure, aortic augmentation index, and precontrast liver computed tomography.

After the study completed, investiators compared the data of interventional groups and placebo groups.

ELIGIBILITY:
Inclusion Criteria:

* TYPE 2 DIABETES MELLITUS PATIENTS WHO CONTROL GLUCOSE BY ORAL ANTIBIABETIC DRUGS OR LIFESTYLE ONLY
* DID NOT CHANGE ANTIDIABETIC DRUG BEFORE THE STUDY FOR 2 MONTHS
* normal physical activity
* 30 to 69 years
* >=6.5% OR <8.0% OF HbA1c

Exclusion Criteria:

* Creatinine>1.5 in men, >1.4 in women
* heavy alcoholics
* who took calcium or vitamin d or anti-osteoporosis drug within 3 months before the study

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2011-12; Primary Completion 2012-10 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
glycemic control | 0, 12week, and 24week
  Investigators checked glycemic control status at the enrollment, 12-week, 24- week by HbA1c

SECONDARY OUTCOMES:
arterial stiffenss | at 0 and 24-week
  central blood pressure brachial-ankle pulse wave velocity aortic augmentation index

OTHER OUTCOMES:
non-alcoholic fatty liver diseases and bone turnover marker | at 0 and 24- week
  precontrast liver computed tomography AST, ALT calcium, PTH, bone specific alkaline phosphatase, serum CTX, calcium

CONTACTS AND LOCATIONS:
Overall Officials: OHKHYUN RYU, PROFESSOR, Principal Investigator — Hallym University Medical Center
Locations (1):
- Chuncheon Sacred Heart Hospital, Chuncheon, Gangwon-do, South Korea

REFERENCES:
- [Background] Breslavsky A, Frand J, Matas Z, Boaz M, Barnea Z, Shargorodsky M. Effect of high doses of vitamin D on arterial properties, adiponectin, leptin and glucose homeostasis in type 2 diabetic patients. Clin Nutr. 2013 Dec;32(6):970-5. doi: 10.1016/j.clnu.2013.01.020. Epub 2013 Feb 27. PMID 23561637